CLINICAL TRIAL: NCT03159299
Title: Yo Puedo! Diabetes Self-Management Education + mHealth in Mexico City
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Yale University (Other)
Collaborators: Universidad Iberoamericana (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Supportive Care
Other Study IDs: 1511016854
Record Dates: First submitted 2017-05-04; First posted 2017-05-18 (Actual); Results first posted 2020-04-27 (Actual); Last update posted 2020-04-27 (Actual); Status verified 2020-04

CONDITIONS: Type 2 Diabetes Mellitus
Keywords: mHealth; Hispanic/Latinos; Diabetes Self-Management Education
MeSH Terms: conditions — Diabetes Mellitus, Type 2 | interventions — Telemedicine

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Yo Puedo (Experimental): This group will receive the modified Yo Puedo + mHealth program.
  Interventions: Behavioral: Yo Puedo + mHealth
- Wait-list Control (No Intervention): This group will not receive the Yo Puedo + mHealth program during the 6 month data collection period, but will be invited to participate in it after data collection has finished.

INTERVENTIONS:
Behavioral: Yo Puedo + mHealth — This intervention is an adapted diabetes self-management education program. Study participants will attend group classes weekly for 6 weeks, and receive daily text messages over 6 months.
  Arms: Yo Puedo

SUMMARY:
The aims of this study are:

1. To translate an evidence-based diabetes self-management education (DSME) program, Yo Puedo!, to the cultural norms, expertise of providers, and systems of care in Seguro Popular clinics in Mexico. The program will be adapted through a collaborative team of diabetes experts in the US and Mexico, Seguro Popular clinic administrators, physicians, nurses and adults with type 2 diabetes (T2D) in Mexico City, Mexico. This will include development and testing of a theory-based mHealth (pictorial text-messaging) component.
2. To evaluate the feasibility (process of implementation, fidelity of sessions, attendance, attrition), acceptability (interviews with nurse, CHW, participants) and preliminary efficacy of Yo Puedo!+mHealth in adults with T2D in Mexico City. A randomized, controlled pilot study design will be used in which 40 adults with T2D are randomized to the Yo Puedo! + mHealth or a wait-list control condition with the hypothesis that clinical [A1C, body mass index (BMI), blood pressure (BP)], T2D self-management, and self-efficacy outcomes will be greater in You Puedo!+mHealth participants compared to the wait-list control condition at 3 and 6 month follow-up. A secondary hypothesis that the Yo Puedo! + mHealth program is feasible and acceptable to adults with T2D and providers and that fidelity of the program will be maintained.

DETAILED DESCRIPTION:
This mixed-method design study will be accomplished in two phases with an interdisciplinary, bi-national collaboration between the Yale School of Nursing, the Yale School of Public Health, the Iberoamericana University in Mexico City, and up to 10 Seguro Popular clinics to evaluate the adapted DSME program for adults with T2D in Mexico City.

Phase 1: While the Yo Puedo! program addresses some of the needs of Mexican adults with type 2 diabetes - interactive health education for low health literacy, Spanish language materials and video novellas, and activities to enhance self-efficacy, the program was developed to address the needs of Latino immigrants in the U.S, who are from different Latin countries. The program needs to be adapted to Mexican adults with respect to personal beliefs about disease causation, cultural health practices, self-care practices of type 2 diabetes, and issues regarding access to care. This aim will be accomplished by using an interpretive and participatory method with a collaborative team of diabetes experts in the US and Mexico, Seguro Popular clinic administrators, physicians, and nurses, and adults with T2D in Mexico City, Mexico. In focus groups and interviews, the study team will explore how the cultural context, family, and health system shape beliefs and practices related to T2D. Access and familiarity with texting technology to identify potential barriers to using a text-messaging mHealth program will also be explored. These results will inform any modifications to the Yo Puedo! curriculum that may need to be made before Phase 2 can begin.

Phase 2: A randomized, controlled pilot study design will be used in which 40 adults with T2D are randomized to the Yo Puedo + mHealth or wait-list control condition with the hypothesis that clinical (A1C, BMI, BP), T2D self-management, and self-efficacy outcomes will be greater in Yo Puedo + mHealth participants compared to the wait-list control condition at 3 and 6 month follow-up. It is also hypothesized that the Yo Puedo + mHealth program is feasible and acceptable to adults with T2D and providers, and that fidelity of the program will be maintained. Those in the control group will be invited to participate in the program after completion of the 6-month data collection. Interviews will be conducted with the nurse, community health worker (CHW), participants, and select clinic personnel to identify barriers, facilitators, and acceptability of the program from multiple perspectives, recognizing the complexity of the health care system. Detailed notes on the process of implementation will be carefully recorded with the purpose of identifying successful and unsuccessful components of the program (positive and negative feedback loops in a complex system).

Setting. The study will be conducted in up to 10 Seguro Popular clinics. These clinics are part of the Social Protection System in Health in Mexico. Individuals who obtain health care at these clinics are covered by public health insurance (Seguro Popular), and the services offered for T2D care include medical visits, referrals to specialists and nutritionist when needed, laboratory testing, and free medicines. The medical visits include medication prescription, blood pressure management, lipid monitoring, and eye/foot care. Laboratory analyses vary from patient to patient but generally includes 3 annual tests of A1C, although other glucose, urine, and lipids tests are also available. Patients with complications are referred to specialized health centers. Evidence suggests that the impact of the Seguro Popular in adults with T2D has been positive.

Interventions. All participants will receive standard T2D care at a Seguro Popular clinic as described above. The wait-list control condition group will receive a handout on T2D self-management and the opportunity to participate in the Yo Puedo! + mHealth program at the completion of 6-month data collection. The Yo Puedo! + mHealth DSME program includes: a) an initial consultation with the nurse to collaboratively determine goals; b) five interactive group-based sessions led by the CHW on T2D self-management that is culturally relevant and at a low health literacy level (Yo Puedo! protocol adapted for Mexican context; c) behavioral support to collaboratively problem-solve barriers to change; and d) empowerment-based strategies to facilitate provider-patient communication. The Yo Puedo! program will be supplemented by 2-way text-messaging capability provided by a web-based platform with privacy and security rules, which allows for automated and personalized messages and a database to store all messages. Automated daily text messages will include messages to promote understanding of T2D self-management, self-efficacy, and adherence to self-management goals. The in-person component will be 6 weeks; daily text messaging will be for 6 months.

ELIGIBILITY:
Inclusion Criteria:

Phase 1:

* For provider interviews/focus groups: administrator or health care provider at Seguro Popular clinic with at least 3 months experience.
* For adult interviews/focus groups: 21-65 years of age and have had T2D for at least one year

Phase 2:

* Age 21-65 years; receiving care for T2D at a Seguro Popular clinic; diagnosed with T2D with A1C >8.0% and duration ≤ 5 years; medically stable and safe to exercise; and have a cell phone (MMS text-messaging will be provided).

Exclusion Criteria:

Phase 2:

* Cognitive impairment, severe untreated clinical depression in the past 6 months, major cardiac event in past 12 months, uncontrolled blood pressure, resting tachycardia, renal failure, severe peripheral neuropathy, treatment of T2D with insulin, and participation in focus groups or interviews.

Ages: 21 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 47 (Actual)
Dates: Start 2017-05-08 (Actual); Primary Completion 2019-04-28 (Actual); Study Completion 2019-06-30 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Robin Whittemore, PhD, Principal Investigator — Yale University
Locations (1):
- Yale School of Nursing, Orange, Connecticut, United States

IPD SHARING:
Plan to Share IPD: Yes
Supporting Information: Study Protocol, SAP
Time Frame: April 2020 - December 2020
Access Criteria: Contact the Principal Investigator

REFERENCES:
- [Derived] Whittemore R, Vilar-Compte M, De La Cerda S, Delvy R, Jeon S, Burrola-Mendez S, Pardo-Carrillo M, Lozano-Marrufo A, Perez-Escamilla R. inverted exclamation markSi, Yo Puedo Vivir Sano con Diabetes! A Self-Management Randomized Controlled Pilot Trial for Low-Income Adults with Type 2 Diabetes in Mexico City. Curr Dev Nutr. 2020 Apr 14;4(5):nzaa074. doi: 10.1093/cdn/nzaa074. eCollection 2020 May. PMID 32368713

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | Yo Puedo | Wait-list Control
Started | 26 | 21
Completed | 24 | 20
Not Completed | 2 | 1

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Yo Puedo | Wait-list Control | Total
Number analyzed (Participants) | 26 | 21 | 47
Age, Continuous [Mean (Standard Deviation); unit: years] | 53.9 (9.2) | 56.8 (8.3) | 55.4 (8.8)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 17 | 14 | 31
  Male | 9 | 7 | 16
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 26 | 21 | 47
  Not Hispanic or Latino | 0 | 0 | 0
  Unknown or Not Reported | 0 | 0 | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0
  Asian | 0 | 0 | 0
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0
  Black or African American | 0 | 0 | 0
  White | 26 | 21 | 47
  More than one race | 0 | 0 | 0
  Unknown or Not Reported | 0 | 0 | 0
Region of Enrollment [Number; unit: participants]
  Mexico | 26 | 21 | 47
Marital Status [Count of Participants; unit: Participants] | 15 | 13 | 28

OUTCOME MEASURES:

1. Primary Outcome: Change in Hemoglobin A1C From Baseline
Description: The change in A1C from baseline to 6 months is the result of the Generalized Linear Mixed Models (GLMM) with an intent-to-treat analysis that was used. HbA1c was measured from finger stick blood sample.
Time Frame: Baseline, 3, 6 months
Population: Intention to treat analysis included all observations for all relevant time points used in the calculation.
Measure: Mean (Standard Deviation); unit: percentage HbA1c
Arm/Group | Yo Puedo | Wait-list Control
Number analyzed (Participants) | 26 | 21
percentage HbA1c
  Change from baseline | -1.76 (0.30) | -0.97 (0.33)
  Baseline | 9.32 (1.44) | 9.09 (1.58)
  3 months | 7.85 (1.40) | 8.76 (1.40)
  6 months | 7.56 (1.50) | 8.05 (1.51)
Statistical Analysis 1: Comparison: Yo Puedo vs Wait-list Control; Test type: Superiority; p < 0.15, Mixed Models Analysis; Mean Difference (Final Values) = 0.11

2. Secondary Outcome: Baseline Systolic and Diastolic Blood Pressure
Description: Systolic and diastolic BP will be measured according to practice standards. Two readings separated by 1 minute will be averaged
Time Frame: Baseline
Reporting Status: Not Posted

3. Secondary Outcome: Change in Baseline Systolic and Diastolic Blood Pressure From Baseline
Description: as for outcome 2
Time Frame: 3 months
Reporting Status: Not Posted

4. Secondary Outcome: Change in Baseline Systolic and Diastolic Blood Pressure From Baseline
Description: as for outcome 2
Time Frame: 6 months
Reporting Status: Not Posted

5. Secondary Outcome: Body Mass Index (BMI)
Description: A calibrated electronic scale will be used to record weight and a wall-based stadiometer will be used to record height. Weight and height will be combined to report BMI in kg/m^2.
Time Frame: Baseline
Reporting Status: Not Posted

6. Secondary Outcome: Change in Body Mass Index (BMI) From Baseline
Description: as for outcome 5
Time Frame: 3 months
Reporting Status: Not Posted

7. Secondary Outcome: Change in Body Mass Index (BMI) From Baseline
Description: as for outcome 5
Time Frame: 6 months
Reporting Status: Not Posted

8. Secondary Outcome: Diabetes Self-management
Description: Measured by the Summary of Diabetes Self-Care Activities questionnaire, a multi-dimensional12-item scale with items on general diet, specific diet, monitoring blood glucose, foot care, and smoking
Time Frame: Baseline
Reporting Status: Not Posted

9. Secondary Outcome: Change in Diabetes Self-management From Baseline
Description: as for outcome 8
Time Frame: 3 months
Reporting Status: Not Posted

10. Secondary Outcome: Change in Diabetes Self-management From Baseline
Description: as for outcome 8
Time Frame: 6 months
Reporting Status: Not Posted

11. Secondary Outcome: Dietary Intake
Description: Dietary intake will be evaluated by a two-day diet history
Time Frame: Baseline
Reporting Status: Not Posted

12. Secondary Outcome: Change in Dietary Intake From Baseline
Description: Dietary intake will be evaluated by a two-day diet history
Time Frame: 3 months
Reporting Status: Not Posted

13. Secondary Outcome: Change in Dietary Intake From Baseline
Description: Dietary intake will be evaluated by a two-day diet history
Time Frame: 6 months
Reporting Status: Not Posted

14. Secondary Outcome: Physical Activity
Description: Physical activity will be measured by accelerometer, using the Actigraph Actigraphy, a 3-axial accelerometer.
Time Frame: Baseline
Reporting Status: Not Posted

15. Secondary Outcome: Change in Physical Activity From Baseline
Description: Physical activity will be measured by accelerometer, using the Actigraph Actigraphy, a 3-axial accelerometer.
Time Frame: 3 months
Reporting Status: Not Posted

16. Secondary Outcome: Change in Physical Activity From Baseline
Description: Physical activity will be measured by accelerometer, using the Actigraph Actigraphy, a 3-axial accelerometer.
Time Frame: 6 months
Reporting Status: Not Posted

17. Secondary Outcome: Diabetes Self-Efficacy
Description: Self-efficacy will be measured by the Stanford Diabetes Self-Efficacy Scale, an 8-item scale specific to T2D self-management self-efficacy.
Time Frame: Baseline
Reporting Status: Not Posted

18. Secondary Outcome: Change in Diabetes Self-Efficacy From Baseline
Description: as for outcome 17
Time Frame: 3 months
Reporting Status: Not Posted

19. Secondary Outcome: Change in Diabetes Self-Efficacy From Baseline
Description: as for outcome 17
Time Frame: 6 months
Reporting Status: Not Posted

20. Other Pre Specified Outcome: Satisfaction With Program
Description: This measure will be used to evaluate the acceptability of the Yo Puedo program. Participants will be given a short survey and interview about their experience and satisfaction with the program.
Time Frame: 6 months
Reporting Status: Not Posted

21. Other Pre Specified Outcome: Rate of Recruitment
Description: Rates of recruitment will be collected by researchers to evaluate feasibility.
Time Frame: through study completion, about 1 year
Reporting Status: Not Posted

22. Other Pre Specified Outcome: Attrition
Description: This will be collected by researchers to evaluate feasibility. The number of participants who do not complete the study interventions and the reasons why will be recorded by study personnel.
Time Frame: through study completion, about 1 year
Reporting Status: Not Posted

23. Other Pre Specified Outcome: Protocol Implementation
Description: This will be collected by researchers to evaluate feasibility. The CHWs will complete a Protocol Implementation Form after each session that documents attendance, length of the session, content of session, protocol implementation, and any deviation from protocol implementation
Time Frame: through study completion, about 1 year
Reporting Status: Not Posted

24. Other Pre Specified Outcome: Fidelity of Yo Puedo Sessions
Description: This will be collected by researchers to evaluate feasibility. A study Co-Investigator will observe 10% of sessions to evaluate fidelity of Yo Puedo sessions.
Time Frame: through study completion, about 1 year
Reporting Status: Not Posted

ADVERSE EVENTS:
Time Frame: Approximately one year
Description: Data were collected on episodes of hypoglycemia or hyperglycemia at data collection times (3 and 6 months). There were 10 minor adverse events of hyperglycemia or hypoglycemia possibly or unrelated to study. There was one major adverse event of hypoglycemia requiring emergency room treatment of participant in the control group, unlikely related to the study. All treatment-related and non-treatment related adverse events are being reported.
Arm/Group | Yo Puedo | Wait-list Control
All-Cause Mortality (participants affected / at risk) | 0/26 | 0/21
Serious Adverse Events (participants affected / at risk) | 0/26 | 1/21
Other Adverse Events (participants affected / at risk) | 8/26 | 2/21
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Yo Puedo (N=26) | Wait-list Control (N=21)
Hypoglycemia (Endocrine disorders) | 0 (0) | 1 (1) — Severe hypoglycemia requiring emergency room treatment
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Yo Puedo (N=26) | Wait-list Control (N=21)
Hypoglycemic (Endocrine disorders) | 5 (5) | 2 (2) — Minor hypoglycemia resolved without medical intervention other than food for hypoglycemia.
hyperglycemia (Endocrine disorders) | 3 (3) | 0 (0) — Minor hyperglycemia resolved without treatment

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2018-10-17): https://cdn.clinicaltrials.gov/large-docs/99/NCT03159299/Prot_SAP_000.pdf